CLINICAL TRIAL: NCT04172181
Title: Multi-center Clinical Study of Cord Blood Stem Cell Transplantation for Severe Combined Immunodeficiency Disease
Brief Title: Multi-center Clinical Study of Cord Blood Stem Cell Transplantation for SCID
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Children's Hospital of Fudan University (Other)
Collaborators: Shanghai Children's Hospital (Other); Children's Hospital of Soochow University (Other); Beijing Children's Hospital (Other); Guangzhou Women and Children's Medical Center (Other); Shenzhen Children's Hospital (Other Government); Wuhan Women and Children's Medical Center (Other); Children's Hospital of Nanjing Medical University (Other); The First Affiliated Hospital of Zhengzhou University (Other)
Responsible Party: Principal Investigator, Xiaowen Zhai, clinical professor, Children's Hospital of Fudan University
Other Study IDs: CPBMT-SCID-2019
Record Dates: First submitted 2019-11-12; First posted 2019-11-21 (Actual); Last update posted 2020-01-28 (Actual); Status verified 2020-01

CONDITIONS: Severe Combined Immunodeficiency Disease
Keywords: cord blood stem cell transplantation; severe combined immunodeficiency disease; primary immunodeficiency
MeSH Terms: conditions — X-Linked Combined Immunodeficiency Diseases; Primary Immunodeficiency Diseases | interventions — Cord Blood Stem Cell Transplantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood sample of every patient will be collected pre and post-transplant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- UCBT-SCID-Case: SCID patients who underwent cord blood stem cell transplantation.The only curative therapy for SCID is allogeneic hematopoietic stem cell transplantation.
  Interventions: Procedure: cord blood stem cell transplantation

INTERVENTIONS:
Procedure: cord blood stem cell transplantation — Unrelated cord blood stem cell selection； Reduced intensity conditioning； GVHD prevention； Infection prevention.

SUMMARY:
Severe combined immunodeficiency (SCID) is a rare disease caused by a group of genetic disorders that leads to early death from recurrent infections in affected children.The only curative therapy for SCID is allogeneic hematopoietic stem cell transplantation.Unrelated umbilical cord blood(UCB) is increasingly used as an alternative to bone marrow.

DETAILED DESCRIPTION:
Severe combined immunodeficiency (SCID) is a rare disease caused by a group of genetic disorders that leads to early death from recurrent infections in affected children.The only curative therapy for SCID is allogeneic hematopoietic stem cell transplantation.Unrelated umbilical cord blood(UCB) is increasingly used as an alternative to bone marrow.The development of NBS in Europe and America has enabled more SCID patients to be diagnosed before symptoms appear, and to enter the normative assessment and intervention procedures as soon as possible. In China SCID has not been included in the NBS program,and there are few units that can diagnose SCID.Patients often delay diagnosis and miss the best period of transplantation. Department of Hematology, Children's Hospital of Fudan University, has used UCBT for the treatment of SCID patients with reduced intensity conditioning(RIC)since 2014.6 of 8 cases were treated with disease-free survival. The encouraging efficacy of these patients suggests that RIC of UCBT may be an effective treatment for SCID patients to urgently hematopoietic stem cell transplantation. The aim of this study is to investigate the efficacy of UCBT in the treatment of SCID, including engraftment rate, disease-free survival rate,overall survival rate and immune reconstitution, and to evaluate transplant-related mortality and complications. All the selected cases are diagnosed as severe combined immunodeficiency disease by immunological function and gene detection. These patients have no matched sibling donors. Their organs function should be normal. The guardian of the patient has the desire and requirement for UCBT and signs the informed consent before treatment. Cord blood stem cell selection:HLA high-resolution detection of patients before transplantation, searching through cord blood stem cell bank, selecting cord blood stem cells that meet the following criteria: HLA-A, B, C, DRB1 high-resolution (genotype) > 6/8matching,total number of nuclear cells >5x10^7/kg.Conditioning:busulfan+ cyclophosphamide.GVHD prevention: tacrolimus (FK506) or cyclosporine A. Infection prevention: Micafungin/caspofungin before engraftment, voriconazole after engraftment to prevent fungi. Ganciclovir is used from the beginning of conditioning to the infusion of cord blood stem cells, and acyclovir is used to prevent virus infection. SMZ prevents Pneumocystis carinii infection after engraftment until half a year after the withdrawal of immunosuppressive agents.

This is a multicenter prospective observational study. Procedure/Surgery: Cord Blood Stem Cell Transplantation Unrelated cord blood stem cell selection: HLA high-resolution detection is performed before transplantation. High-resolution (genotype) matching of HLA-A, B, C and DRB1 was selected. The total number of nuclear cells is more than 5*107/kg.

Reduced intensity conditioning : Busulphan 3.2mg/kg per day in divided doses for 3 days(total dose 9.6 mg/kg) and cyclophosphamide 50 mg/kg for 2 days (total dose 100 mg/kg).

GVHD prevention: tacrolimus (FK506) 0.1 mg/kg/day, started 4 days before transplantation, is taken orally twice, and the blood concentration is monitored to maintain the concentration at 5-10 ng/ml. If the patient does not have a GVHD transplant +100 days after the slow reduction, until the transplant 6 months after the withdrawal.

Infection prevention: Micafungin/caspofungin before engraftment, voriconazole after engraftment to prevent fungi. Ganciclovir is used from the beginning of pretreatment to the beginning of reinfusion, and acyclovir is used to prevent virus infection until immunosuppressive agents are discontinued after reinfusion. SMZ prevents Pneumocystis carinii infection after engraftment.

ELIGIBILITY:
Inclusion Criteria:

1. All patients were diagnosed as severe combined immunodeficiency disease by immunological function and genetic diagnosis center.
2. Patients have no HLA-matched related donor.
3. Each organ functions normally and conforms the following inspection criteria:

Liver function ALT, AST ≤ 10 times the upper limit of normal value, TBIL ≤ 5 times the upper limit of normal value.

Renal function BUN, Cr ≤ 1.25 times the upper limit of normal value. ECG, cardiac examination normal

Exclusion Criteria:

1. Patients have any contraindications to hematopoietic stem cell transplantation.
2. Patients have other serious diseases, such as serious damage to vital organ function: respiratory failure, cardiac insufficiency, decompensated liver dysfunction, renal insufficiency, uncontrollable infection, etc.
3. The patient is undergoing other drug clinical research.
4. At the same time suffering from other serious acute or chronic physical or mental illness, or laboratory abnormalities, may affect patient safety and compliance, affecting informed consent, research participation, follow-up or interpretation of results.

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients were diagnosed as severe combined immunodeficiency disease by immunological function and genetic diagnosis center.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2019-12-01 (Actual); Primary Completion 2022-10-31 (Estimated); Study Completion 2023-10-31 (Estimated)

PRIMARY OUTCOMES:
Overall survival rate | 3 years after transplantation
  Overall survival is defined as the survival status of patients by the end of 3 years after the transplanting, coded as 1 for dead and 0 for survive.

SECONDARY OUTCOMES:
Disease free survival rate | 3 years after transplantation
  Disease free survival is defined as the survival status of patients by the end of the third year after transplantation. Disease free survival is defined as survive without conditions including engraftment failure and death caused by any reasons. The variable is coded as 0 for disease free survive, and 1 for all conditions other than the defined status of "0".
Successful engraftment | 3 years after transplantation
  The event of successful engraftment is defined as Neutrophil count ≥ 0.5×10^9/L for continuous 3 days and platelet count ≥ 20×10^9/L for continuous 7 days without transfusion. It is coded as 1.
Immune reconstitution | 3 years after transplantation
  Immune reconstitution is including T-cell and B-cell reconstitution.The variable would be coded as 1 if any of these two cells had been reconstituted while 0 for none. T-cell reconstitution is defined as meeting these criteria: CD3+ cell count > 1000 per cubic millimeter, and CD4+ cell count > 500 per cubic millimeter. B-cell reconstitution is defined as independence from Ig-replacement therapy.

OTHER OUTCOMES:
The occurrence of adverse events (AE) | 3 years after transplantation
  The adverse events (AE) is a composite variable including liver and kidney function damage, nausea, vomiting, arrhythmia and dyspnea. The variable would be coded as 1 if any of these events occurs after transplantation for 3 years while 0 for none . These adverse events would be measured by assessment scale method according to NCI CTC AE v4.0 classification standard.
The occurrence of graft-versus-host disease (GVHD) | 3 years after transplantation
  Acute and chronic GVHD is measured and graded as per standardised criteria.
Transplant-related mortality | 3 years after transplantation
  Transplant-related mortality (TRM)included mortality from any cause other than as a result of the underlying primary immunodeficiency up to day +100 post neutrophil engraftment.
The occurrence of transplant-related complications except GVHD | 3 years after transplantation
  Transplant-related complications include infections, hepatic venous occlusion disease, hemorrhagic cystitis, capillary leakage syndrome, thrombotic microangiopathy, post-transplantation lymphoproliferative disease, idiopathic pneumonia syndrome and obstructive bronchiolitis, which are diagnosed according to the relevant diagnosis standards of each disease.

CONTACTS AND LOCATIONS:
Overall Officials: jiang hui, master, Study Director — Shanghai Children's Hospital; hu shaoyan, PhD, Study Director — Children's Hospital of Soochow University; qin maoquan, master, Study Director — Beijing Children's Hospital; jiang hua, PhD, Study Director — Guangzhou Women and Children's Medical Center; liu sixi, master, Study Director — Shenzhen Children's Hospital; xiong hao, PhD, Study Director — Wuhan Women and Children's Medical Center; fang yongjun, PhD, Study Director — Children's Hospital of Nanjing Medical University; wang dao, PhD, Study Director — The First Affiliated Hospital of Zhengzhou University
Locations (1):
- Children's Hospital of Fudan University, Shanghai, Minhang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] van der Burg M, Gennery AR. Educational paper. The expanding clinical and immunological spectrum of severe combined immunodeficiency. Eur J Pediatr. 2011 May;170(5):561-71. doi: 10.1007/s00431-011-1452-3. Epub 2011 Apr 9. PMID 21479529
- [Result] Gaspar HB, Qasim W, Davies EG, Rao K, Amrolia PJ, Veys P. How I treat severe combined immunodeficiency. Blood. 2013 Nov 28;122(23):3749-58. doi: 10.1182/blood-2013-02-380105. Epub 2013 Oct 10. PMID 24113871
- [Result] Pai SY, Logan BR, Griffith LM, Buckley RH, Parrott RE, Dvorak CC, Kapoor N, Hanson IC, Filipovich AH, Jyonouchi S, Sullivan KE, Small TN, Burroughs L, Skoda-Smith S, Haight AE, Grizzle A, Pulsipher MA, Chan KW, Fuleihan RL, Haddad E, Loechelt B, Aquino VM, Gillio A, Davis J, Knutsen A, Smith AR, Moore TB, Schroeder ML, Goldman FD, Connelly JA, Porteus MH, Xiang Q, Shearer WT, Fleisher TA, Kohn DB, Puck JM, Notarangelo LD, Cowan MJ, O'Reilly RJ. Transplantation outcomes for severe combined immunodeficiency, 2000-2009. N Engl J Med. 2014 Jul 31;371(5):434-46. doi: 10.1056/NEJMoa1401177. PMID 25075835
- [Result] Chan K, Puck JM. Development of population-based newborn screening for severe combined immunodeficiency. J Allergy Clin Immunol. 2005 Feb;115(2):391-8. doi: 10.1016/j.jaci.2004.10.012. PMID 15696101
- [Result] Routes JM, Grossman WJ, Verbsky J, Laessig RH, Hoffman GL, Brokopp CD, Baker MW. Statewide newborn screening for severe T-cell lymphopenia. JAMA. 2009 Dec 9;302(22):2465-70. doi: 10.1001/jama.2009.1806. PMID 19996402
- [Result] Gatti RA, Meuwissen HJ, Allen HD, Hong R, Good RA. Immunological reconstitution of sex-linked lymphopenic immunological deficiency. Lancet. 1968 Dec 28;2(7583):1366-9. doi: 10.1016/s0140-6736(68)92673-1. No abstract available. PMID 4177932
- [Result] Antoine C, Muller S, Cant A, Cavazzana-Calvo M, Veys P, Vossen J, Fasth A, Heilmann C, Wulffraat N, Seger R, Blanche S, Friedrich W, Abinun M, Davies G, Bredius R, Schulz A, Landais P, Fischer A; European Group for Blood and Marrow Transplantation; European Society for Immunodeficiency. Long-term survival and transplantation of haemopoietic stem cells for immunodeficiencies: report of the European experience 1968-99. Lancet. 2003 Feb 15;361(9357):553-60. doi: 10.1016/s0140-6736(03)12513-5. PMID 12598139
- [Result] Fernandes JF, Rocha V, Labopin M, Neven B, Moshous D, Gennery AR, Friedrich W, Porta F, Diaz de Heredia C, Wall D, Bertrand Y, Veys P, Slatter M, Schulz A, Chan KW, Grimley M, Ayas M, Gungor T, Ebell W, Bonfim C, Kalwak K, Taupin P, Blanche S, Gaspar HB, Landais P, Fischer A, Gluckman E, Cavazzana-Calvo M; Eurocord and Inborn Errors Working Party of European Group for Blood and Marrow Transplantation. Transplantation in patients with SCID: mismatched related stem cells or unrelated cord blood? Blood. 2012 Mar 22;119(12):2949-55. doi: 10.1182/blood-2011-06-363572. Epub 2012 Feb 3. PMID 22308292
- [Result] Chiesa R, Gilmour K, Qasim W, Adams S, Worth AJ, Zhan H, Montiel-Equihua CA, Derniame S, Cale C, Rao K, Hiwarkar P, Hough R, Saudemont A, Fahrenkrog CS, Goulden N, Amrolia PJ, Veys P. Omission of in vivo T-cell depletion promotes rapid expansion of naive CD4+ cord blood lymphocytes and restores adaptive immunity within 2 months after unrelated cord blood transplant. Br J Haematol. 2012 Mar;156(5):656-66. doi: 10.1111/j.1365-2141.2011.08994.x. Epub 2012 Jan 9. PMID 22224700
- [Result] Gennery AR, Slatter MA, Grandin L, Taupin P, Cant AJ, Veys P, Amrolia PJ, Gaspar HB, Davies EG, Friedrich W, Hoenig M, Notarangelo LD, Mazzolari E, Porta F, Bredius RG, Lankester AC, Wulffraat NM, Seger R, Gungor T, Fasth A, Sedlacek P, Neven B, Blanche S, Fischer A, Cavazzana-Calvo M, Landais P; Inborn Errors Working Party of the European Group for Blood and Marrow Transplantation; European Society for Immunodeficiency. Transplantation of hematopoietic stem cells and long-term survival for primary immunodeficiencies in Europe: entering a new century, do we do better? J Allergy Clin Immunol. 2010 Sep;126(3):602-10.e1-11. doi: 10.1016/j.jaci.2010.06.015. Epub 2010 Jul 31. PMID 20673987
- [Result] Grunebaum E, Mazzolari E, Porta F, Dallera D, Atkinson A, Reid B, Notarangelo LD, Roifman CM. Bone marrow transplantation for severe combined immune deficiency. JAMA. 2006 Feb 1;295(5):508-18. doi: 10.1001/jama.295.5.508. PMID 16449616
- [Result] de la Morena MT, Nelson RP Jr. Recent advances in transplantation for primary immune deficiency diseases: a comprehensive review. Clin Rev Allergy Immunol. 2014 Apr;46(2):131-44. doi: 10.1007/s12016-013-8379-6. PMID 23832379
- [Result] Castillo N, Garcia-Cadenas I, Barba P, Canals C, Diaz-Heredia C, Martino R, Ferra C, Badell I, Elorza I, Sierra J, Valcarcel D, Querol S. Early and Long-Term Impaired T Lymphocyte Immune Reconstitution after Cord Blood Transplantation with Antithymocyte Globulin. Biol Blood Marrow Transplant. 2017 Mar;23(3):491-497. doi: 10.1016/j.bbmt.2016.11.014. Epub 2016 Nov 22. PMID 27888015
- [Result] Williams KM, Hakim FT, Gress RE. T cell immune reconstitution following lymphodepletion. Semin Immunol. 2007 Oct;19(5):318-30. doi: 10.1016/j.smim.2007.10.004. Epub 2007 Nov 19. PMID 18023361
- [Result] Walker CM, van Burik JA, De For TE, Weisdorf DJ. Cytomegalovirus infection after allogeneic transplantation: comparison of cord blood with peripheral blood and marrow graft sources. Biol Blood Marrow Transplant. 2007 Sep;13(9):1106-15. doi: 10.1016/j.bbmt.2007.06.006. PMID 17697973
- [Result] Beck JC, Wagner JE, DeFor TE, Brunstein CG, Schleiss MR, Young JA, Weisdorf DH, Cooley S, Miller JS, Verneris MR. Impact of cytomegalovirus (CMV) reactivation after umbilical cord blood transplantation. Biol Blood Marrow Transplant. 2010 Feb;16(2):215-22. doi: 10.1016/j.bbmt.2009.09.019. Epub 2009 Sep 26. PMID 19786112
- [Result] Szabolcs P, Niedzwiecki D. Immune reconstitution in children after unrelated cord blood transplantation. Biol Blood Marrow Transplant. 2008 Jan;14(1 Suppl 1):66-72. doi: 10.1016/j.bbmt.2007.10.016. Erratum In: Biol Blood Marrow Transplant. 2008 Nov;14(11):1317-8. PMID 18162223
- [Result] Uhlin M, Sairafi D, Berglund S, Thunberg S, Gertow J, Ringden O, Uzunel M, Remberger M, Mattsson J. Mesenchymal stem cells inhibit thymic reconstitution after allogeneic cord blood transplantation. Stem Cells Dev. 2012 Jun 10;21(9):1409-17. doi: 10.1089/scd.2011.0310. Epub 2011 Oct 12. PMID 21861757
- [Result] Krenger W, Hollander GA. The immunopathology of thymic GVHD. Semin Immunopathol. 2008 Dec;30(4):439-56. doi: 10.1007/s00281-008-0131-6. Epub 2008 Oct 31. PMID 18974988
- [Result] Weinberg K, Blazar BR, Wagner JE, Agura E, Hill BJ, Smogorzewska M, Koup RA, Betts MR, Collins RH, Douek DC. Factors affecting thymic function after allogeneic hematopoietic stem cell transplantation. Blood. 2001 Mar 1;97(5):1458-66. doi: 10.1182/blood.v97.5.1458. PMID 11222394
- [Result] Chung B, Barbara-Burnham L, Barsky L, Weinberg K. Radiosensitivity of thymic interleukin-7 production and thymopoiesis after bone marrow transplantation. Blood. 2001 Sep 1;98(5):1601-6. doi: 10.1182/blood.v98.5.1601. PMID 11520813
- [Result] Jimenez M, Martinez C, Ercilla G, Carreras E, Urbano-Ispizua A, Aymerich M, Villamor N, Amezaga N, Rovira M, Fernandez-Aviles F, Gaya A, Martino R, Sierra J, Montserrat E. Reduced-intensity conditioning regimen preserves thymic function in the early period after hematopoietic stem cell transplantation. Exp Hematol. 2005 Oct;33(10):1240-8. doi: 10.1016/j.exphem.2005.06.016. PMID 16219547